CLINICAL TRIAL: NCT03683784
Title: Prevalence of Type 2 Diabetes in Fayoum Governorate
Brief Title: Type 2 Diabetes in Fayoum
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelkawi Hammad, Lecturer of internal medicine, Fayoum University
Other Study IDs: D75
Record Dates: First submitted 2018-09-24; First posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Males: Male diabetics or male subjects proved to be diabetics
- Female: Female diabetics or male subjects proved to be diabetics

SUMMARY:
study the prevalence of type II diabetes mellitus, prevalence of newly diagnosed type II diabetic patients

DETAILED DESCRIPTION:
study the prevalence of type II diabetes mellitus, prevalence of newly diagnosed type II diabetic patients, status of glycemic control and associated risk factors and complications of diabetes among population of Fayoum governorate

ELIGIBILITY:
Inclusion Criteria:

* community sample as obese persons,family history of diabetes,diabetics,hypertensives,dyslipidemics

Exclusion Criteria:

* subjects known to have:chronic liver disease,CKD,Cushing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: obese persons,dyslipidemics ,apparently healthy individuals
Sampling Method: Probability Sample
Enrollment: 3500 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of diabetes in Fayoum | 11 months
  Prevalence of diabetes in Fayoum governorate

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Hammad, MD, Study Director — Fayoum University

IPD SHARING:
Plan to Share IPD: Undecided
Probably will